CLINICAL TRIAL: NCT04294680
Title: Prospective, Randomized, Controlled Trial of an Opiate Sparing Protocol Versus Standard Opiate-Based Protocol Following Shoulder Arthroplasty
Brief Title: Opiate Sparing Versus Opiate Based Following Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Tyler J. Brolin, Principal Investigator, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BMH 19-29
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Surgery
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Opiate Sparing (Experimental): Cryotherapy one hour daily four times per day for two weeks postoperative Acetaminophen 1000 milligrams every six hours by mouth for fourteen days postoperative Gabapentin 100 milligrams three times per day by mouth for thirty days postoperative Celecoxib 100 milligrams two times per day by mouth for thirty days postoperative Esomeproazole 20 milligrams daily by mouth for thirty days postoperative Ondansetron 4 milligrams every eight hours by mouth as needed for nausea and/or vomiting for fourteen days postoperative Oxycodone 5 milligrams every six hours by mouth as needed for uncontrolled pain for fourteen days postoperative
  Interventions: Device: Cryotherapy
- Opiate Based (No Intervention): Oxycodone 5 to 10 milligrams every four to six hours by mouth as needed for pain for fourteen days postoperative Acetaminophen 1000 milligrams every six hours by mouth for fourteen days postoperative Gabapentin 100 milligrams three times per day by mouth for thirty days postoperative Celecoxib 100 milligrams two times per day by mouth for thirty days postoperative Esomeprazole 20 milligrams daily by mouth for thirty days postoperative Ondansetron 4 milligrams every eight hours by mouth as needed for nausea and/or vomiting for fourteen days postoperative

INTERVENTIONS:
Device: Cryotherapy — see opiate sparing description
  Arms: Opiate Sparing

SUMMARY:
To investigate the difference between an opiate sparing pain management protocol versus a standard opiate-based protocol following shoulder arthroplasty in the ninety day postoperative period regarding visual analog scores and oral morphine equivalents.

DETAILED DESCRIPTION:
This is a single center, investigator initiated, prospective, randomized, controlled trial conducted among patients who have given voluntary consent to participate. Participation will last until the completion of the twelve weeks standard of care follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Primary shoulder arthroplasty
* 18-85 years of age
* Body Mass Index greater than or equal to 45
* Willing and able to provide written informed consent
* Willing and able to cooperative in the required postoperative therapy
* Willing and able to complete scheduled follow-up evaluations
* Fluent in verbal and written English

Exclusion Criteria:

* Less than 18 years or over 85 years of age
* Unable to provide written informed consent, cooperate with postoperative therapy, or complete follow-up evaluations
* Known sensitivity, allergy, or intolerance to medications with protocols
* Renal disease as defined by active or impending dialysis within six months or kidney transplant
* Concomitant ipsilateral upper extremity injury or condition other than shoulder that compromises function
* Chronic pain syndrome
* Five consecutive days of opiate use with the previous ninety days
* Worker's compensation claim
* Women who are pregnant, planning to become to become pregnant, or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Brolin, MD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opiate Sparing | Opiate Based
Started | 39 | 43
Received Allocated Intervention | 37 (2 patients withdrew consent prior to surgery) | 42 (1 patient withdrew consent before surgery)
Completed | 36 (1 patient was excluded from analysis due to having follow-up visits completed outside of window) | 42
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Follow-up visits completed outside of window | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opiate Sparing | Opiate Based | Total
Number analyzed (Participants) | 36 | 42 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (6.6) | 72.4 (5.4) | 72.24 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 20 | 27 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Race | 34 | 40 | 74
  Other Race | 2 | 2 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (4.1) | 30.2 (6.3) | 30.36 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Score (VAS) at Week 2
Description: The Visual Analog Score (VAS) is a a validated patient reported pain score with possible range from zero (no pain) to ten (worst possible pain).
Time Frame: postoperative day fourteen (two weeks)
Population: All patients that completed surgery, received their assigned intervention, and completed all follow-up visits within the study window
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opiate Sparing | Opiate Based
Number analyzed (Participants) | 36 | 42
score on a scale | 1.4 (1.7) | 1.8 (2.3)

2. Secondary Outcome: Number of Opioid Pain Pills Taken
Description: The total number of opioid pain pills consumed from post-operative day 1 to Week 12
Time Frame: Post-operative Day 1 through 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: opioid pain pills
Arm/Group | Opiate Sparing | Opiate Based
Number analyzed (Participants) | 36 | 42
opioid pain pills | 4.3 (11.9) | 17.0 (19.6)

ADVERSE EVENTS:
Time Frame: Adverse events, postoperative complications, readmissions, and reoperations were recorded from day of surgery through week 12
Arm/Group | Opiate Sparing | Opiate Based
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/42
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/42
Other Adverse Events (participants affected / at risk) | 2/36 | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opiate Sparing (N=36) | Opiate Based (N=42)
Periprosthetic Fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Acromial Stress Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04294680/Prot_SAP_000.pdf